CLINICAL TRIAL: NCT04824794
Title: An Open-Label, Multicenter, Phase 1/2 Trial of GEN3014 (HexaBody®-CD38) in Relapsed or Refractory Multiple Myeloma and Other Hematologic Malignancies
Brief Title: GEN3014 Trial in Relapsed or Refractory Hematologic Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The sponsor has decided to discontinue further development of GEN3014 after a comprehensive review of the data, market landscape, and strategic priorities.
Sponsor: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCT3014-01; 2020-003781-40 (EudraCT Number); NL75422.056.21 (Registry Identifier: The Netherlands CCMO); 2023-507086-26-00 (EU CTIS Number)
Record Dates: First submitted 2021-03-09; First posted 2021-04-01 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Relapsed or Refractory Multiple Myeloma (RRMM); Diffuse Large B Cell Lymphoma (DLBCL); Acute Myeloid Leukemia (AML)
Keywords: Hexabody®; Anti-CD38; monoclonal antibody
MeSH Terms: conditions — Recurrence; Multiple Myeloma; Lymphoma, Large B-Cell, Diffuse; Leukemia, Myeloid, Acute | interventions — daratumumab

STUDY DESIGN:
Intervention Model Description: Dose escalation part is sequential while the expansion Part A cohorts are parallel. Expansion Part B is sequential to Expansion Part A RRMM cohort. In Expansion Part B, participants with RRMM are randomized (1:1) to treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GEN3014 (Experimental): Experimental: GEN3014 Participants in Dose Escalation phase with
  * RRMM
  * R/R AML
  Participants in Expansion Part A with
  * RRMM (anti-CD38 mAb-naïve)
  * RRMM (anti-CD38 mAb-refractory)
  * R/R DLBCL
  * R/R AML
  Participants in Expansion Part B with
  • RRMM (anti-CD38 mAb-naïve)
  Interventions: Biological: GEN3014
- Daratumumab (Active Comparator): Participants in Expansion Part B with
  - RRMM (anti-CD38 mAb-naïve)
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Biological: GEN3014 — GEN3014 is administered by IV infusion.
  Other Names: HexaBody®-CD38
  Arms: GEN3014
Drug: Daratumumab — Daratumumab is administered by SC injections.
  Other Names: DARZALEX FASPRO®
  Arms: Daratumumab

SUMMARY:
The drug that will be investigated in the study is an antibody, GEN3014. Since this is the first study of GEN3014 in humans, the main purpose is to evaluate safety. In addition to safety, the study will determine the recommended GEN3014 dose to be tested in a larger group of participants and assess preliminary clinical activity of GEN3014. GEN3014 will be studied in relapsed (disease has returned) or refractory (resistant to treatment) multiple myeloma (also known as RRMM) and other blood cancers. The study consists of 3 parts:

1. The Dose Escalation will test increasing doses of GEN3014 to identify a safe dose level to be tested in the other two parts.
2. Expansion Part A will further test the GEN3014 dose determined from the Dose Escalation.
3. Expansion Part B will compare intravenous (IV) GEN3014 with the subcutaneous (SC) daratumumab in ex-US countries.

Participants will receive either GEN3014 into the vein or daratumumab under the skin; none will be given placebo. The study duration will be different for the individual participants. Overall, the study may be ongoing up to 5 years after the last participant's first treatment.

DETAILED DESCRIPTION:
This trial will be conducted in 3 parts: Dose Escalation (phase 1), Expansion Parts, A and B (phase 2).

In the dose escalation phase GEN3014 will be evaluated in RRMM and relapsed and refractory acute myeloid leukemia (R/R AML). The participants will receive GEN3014 administered at various dose levels in 28-day cycles. Dose Limiting Toxicities (DLTs) will be assessed during the first treatment cycle and the Maximum Tolerated Dose (MTD) and/or Recommended phase 2 dose (RP2D) will be determined.

In Expansion Part A, GEN3014 will be further evaluated in 4 cohorts: anti-CD38 monoclonal antibody (mAb)-naive RRMM, anti-CD38 mAb-refractory RRMM, relapsed or refractory diffuse large B-cell lymphoma (R/R DLBCL), and R/R AML at the RP2D identified from the Dose Escalation. In Expansion Part B, GEN3014 IV will be compared to daratumumab SC, head-to-head (H2H) to evaluate whether GEN3014 may be more potent in anti-CD38 mAb-naïve RRMM participants.

ELIGIBILITY:
Key Inclusion Criteria

* Must have fresh bone marrow samples collected at Screening for RRMM, R/R AML, and R/R DLBCL with suspected bone marrow involvement.
* Dose Escalation phase, Expansion Part A (for MM and AML) and Expansion Part B- Eastern Cooperative Oncology Group (ECOG) performance status (PS) score 0, 1, or 2. Expansion Part A (for DLBCL): ECOG PS 0 or 1.
* Has acceptable laboratory test results during the Screening period.
* A woman of reproductive potential must agree to use adequate contraception during the trial and for 12 months after the last GEN3014 or daratumumab SC administration.
* A woman of childbearing potential must have a negative serum beta-human chorionic gonadotropin (β-hCG) at Screening and additionally, for Expansion Part B, within 72 hours of the first dose of study treatment prior to dosing.
* A woman must agree not to donate eggs (ova, oocytes) for assisted reproduction during the trial and for 12 months after receiving the last dose of GEN3014 or daratumumab SC.
* A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control and all men must not donate sperm during the trial and for 12 months after receiving the last dose of GEN3014 or daratumumab SC.

Specific for RRMM:

* Must have documented multiple myeloma as defined by the criteria below and have evidence of disease progression on the most recent prior treatment regimen based on IMWG criteria:

  * Prior documentation of monoclonal plasma cells in the bone marrow ≥10% or presence of a biopsy-proven plasmacytoma and,
  * Measurable disease at baseline as defined by any of the following:

    * Immunoglobulin (Ig) G, IgA, IgD, or IgM myeloma: Serum M-protein level ≥0.5 g/dL (≥5 g/L) or urine M protein level ≥200 mg/24 hours or,
    * Light chain myeloma: Serum Ig free light chain (FLC) ≥10 mg/dL and abnormal serum Ig kappa lambda FLC ratio.

Note: Participants with RRMM must have exhausted standard therapies, at the investigator's discretion.

* For anti-CD38 mAb-naive RRMM Cohort: Participant received at least 3 prior lines of therapy including a proteasome inhibitor (PI) and an immunomodulatory imide drug (IMiD) in any order, or is double refractory to a PI and an IMiD; or participant received ≥ 2 prior lines of therapy if 1 of those lines included a combination of PI and IMiD. Note: Participants should not have received any anti-CD38 antibody.
* Anti-CD38 mAb-naive RRMM participants will be enrolled from ex-US countries.
* Dose Escalation phase - For anti-CD38 mAb-treated RRMM Cohort: Participant has received at least 2 prior lines of therapy and must have discontinued daratumumab or isatuximab for at least 4 weeks prior to the first dose of GEN3014. Note: Participants should not have received any other anti-CD38 antibody except daratumumab or isatuximab.

Specific for R/R AML:

* Relapsed or refractory AML, both de novo or secondary; must have failed all conventional therapy. Acute promyelocytic leukemia (APL) is excluded from this trial. Note: Relapse is defined by BM blasts ≥5% in participants who have been in CR previously, or reappearance of blasts in the blood, or development of extramedullary AML. Refractory is defined as not being able to achieve a CR after the initial therapy.
* Participant with relapsed AML who received at least 2 prior therapies for AML with the exception of hydroxyurea.
* Participant with refractory AML who received at least 1 prior line of therapy for AML with the exception of hydroxyurea.
* Participant's life expectancy at Screening is judged to be at least 3 months.

Specific for DLBCL:

* Expansion phase: Relapsed or refractory DLBCL, both de novo or histologically transformed. Participants with R/R DLBCL must have exhausted standard therapies, at the investigator's discretion.
* Expansion phase: Received at least 2 prior lines of systemic therapy, with 1 being a CD20-containing chemoimmunotherapy.
* Expansion phase: Have at least 1 measurable site of disease as per Lugano criteria.
* Expansion phase: Must have available archival or fresh tumor tissue or both to submit to a central laboratory for CD38 assay.

Key Exclusion Criteria

* Prior treatment with any CD38-directed therapies (eg, daratumumab, isatuximab, CD38 chimeric antigen receptor T cell (CAR-T), bispecific antibody (Ab)) in anti-CD38 mAb-naive RRMM Cohort. Note: Prior daratumumab or isatuximab exposure is allowed for anti-CD38 mAb-treated RRMM participants in the Dose Escalation and anti-CD38 mAb-refractory RRMM Cohort in the Expansion Part A.
* Treatment with an anti-cancer agent, chemotherapy, radiation therapy, or major surgery within 2 weeks prior to the first dose of study treatment (Dose Escalation and Expansion Part A) or randomization (Expansion Part B).
* Treatment with an investigational drug within 4 weeks or 5 half-lives, whichever is shorter, prior to the first dose of study treatment (Dose Escalation and Expansion Part A) or randomization (Expansion Part B).
* Cumulative dose of corticosteroids more than the equivalent of ≥140 mg of prednisone within 2-week period before the first dose of study treatment (Dose Escalation and Expansion Part A) or maximum cumulative dose of dexamethasone 160 mg within 28 days of randomization (Expansion Part B).
* Has clinically significant cardiac disease.
* Toxicities from previous anti-cancer therapies have not resolved to baseline levels or to Grade 1 or less except for alopecia and peripheral neuropathy.
* Primary central nervous system (CNS) tumor or known CNS involvement at Screening.
* Has known history/positive serology for hepatitis B.
* Known medical history or ongoing hepatitis C infection that has not been cured.
* Known history of seropositivity of human immunodeficiency virus (HIV) (Dose Escalation and Expansion Part A) or to be positive for HIV with details in the protocol (Expansion Part B).
* Currently receiving any other investigational agents.
* A woman who is pregnant or breast-feeding, or who is planning to become pregnant while enrolled in this trial or within 12 months after the last dose of study treatment.
* A man who plans to father a child while enrolled in this trial or within 12 months after the last dose of study treatment.

Specific Exclusion Criteria for RRMM:

* Prior allogeneic hematopoietic stem cell transplant (HSCT).
* Autologous HSCT within 3 months of the first dose of GEN3014.

Specific Exclusion Criteria for R/R AML:

* <5% blasts in blood or bone marrow at Screening.
* White blood cell (WBC) counts ≥50,000/microliter (μL) in peripheral blood that cannot be controlled by hydroxyurea prior to the first dose of GEN3014.
* Prior autologous HSCT.
* Allogenic HSCT within 3 months of the first dose of GEN3014.
* Active graft-versus-host-disease requiring immunosuppressive treatment. Any immunosuppressive medication (eg, calcineurin inhibitors) must be stopped ≥4 weeks prior to the first dose of GEN3014.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Dose Escalation: Number of Participants with Dose Limiting Toxicities (DLTs) | Up to 28 days during the first cycle (cycle =28 days)
  To determine the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) to be studied in the Expansion part. DLT will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.
Dose Escalation: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From first dose until the end of the safety follow-up period (30 days after last dose; up to 8 years)
Expansion Part A: Objective Response Rate (ORR) of GEN3014 | Up to 8 years
  ORR is defined as the percentage of participants with a partial response (PR), or better based on International Myeloma Working Group (IMWG) criteria for MM participants, based on Lugano criteria for DLBCL participants, and based on International Working Group (IWG) response criteria for AML participants.
Expansion Part B: Objective Response Rate (ORR) of GEN3014 IV vs Daratumumab SC in Anti-CD38 mAb-naive RRMM Participants | Up to 8 years
  ORR is defined as the percentage of participants with a PR, or better based on IMWG criteria.

SECONDARY OUTCOMES:
Dose Escalation: Maximum (peak) Plasma Concentration (Cmax) of GEN3014 | Predose and postdose at multiple timepoints up to Cycle 6 (Cycle length=28 days); Pre-dose and 5 minutes post end of infusion from Cycle 7 and beyond (Up to 8 years)
Dose Escalation: Pre-dose (trough) Concentrations (Ctrough) of GEN3014 | Predose and postdose at multiple timepoints of each Cycle (Cycle length=28 days) (Up to 8 years)
Dose Escalation: Area Under the Concentration Time Curve From Zero to Last Quantifiable Sample (AUC0-last) | Predose and postdose at multiple timepoints up to Cycle 6 (Cycle length=28 days); Pre-dose and 5 minutes post end of infusion from Cycle 7 and beyond (Up to 8 years)
Dose Escalation: Area Under the Concentration Time Curve From Zero to 168 hours (AUC0-168 h) | Predose and postdose at multiple timepoints up to Cycle 6 (Cycle length=28 days); Pre-dose and 5 minutes post end of infusion from Cycle 7 and beyond (Up to 8 years)
Dose Escalation: Number of Participants with Anti-Drug Antibody (ADA) of GEN3014 | From first dose until treatment discontinuation (Up to 8 years)
Dose Escalation: Objective Response Rate (ORR) of GEN3014 | Up to 8 years
  ORR is defined as the percentage of participants with a PR or better based on IMWG criteria for MM participants and based on IWG response criteria for AML participants.
Dose Escalation: Clinical Benefit Rate (CBR) of GEN3014 | Up to 8 years
  CBR was determined by the investigator according to the IMWG response criteria for MM participants.
Dose Escalation: Duration of Response (DOR) of GEN3014 | Up to 8 years
  DOR is defined as time from first response (PR or better) to time of disease progression or death (due to any cause), whichever comes first based on IMWG criteria for MM participants and based on IWG response criteria for AML participants.
Dose Escalation: Time-to-response (TTR) of GEN3014 | Up to 8 years
  TTR is defined as the time from date of first dose to time of response (PR or better) based on IMWG criteria for MM participants and based on IWG response criteria for AML participants.
Dose Escalation: Progression-free survival (PFS) of GEN3014 | Up to 8 years
  PFS is defined as the time from the date of the first dose to the date of progression or death (due to any cause), whichever comes first based on IMWG criteria for MM participants and based on IWG response criteria for AML participants.
Dose Escalation: Overall Survival (OS) of GEN3014 | Up to 8 years
  OS is defined as the time from the date of first dose to the date of death due to any cause.
Expansion Part A: Clinical Benefit Rate (CBR) of GEN3014 | Up to 8 years
  CBR was determined by the investigator according to the IMWG response criteria for MM participants.
Expansion Part A: Duration of Response (DOR) of GEN3014 | Up to 8 years
  DOR is defined as time from first response (PR or better) to time of disease progression or death (due to any cause), whichever comes first based on IMWG criteria for MM participants, based on Lugano criteria for DLBCL participants, and based on IWG response criteria for AML participants.
Expansion Part A: Time-to-response (TTR) of GEN3014 | Up to 8 years
  TTR is defined as the time from date of first dose to time of response (PR or better) for MM participants, based on Lugano criteria for DLBCL participants, and based on IWG response criteria for AML participants.
Expansion Part A: Progression-free survival (PFS) of GEN3014 | Up to 8 years
  PFS is defined as the time from the date of the first dose to the date of progression or death (due to any cause), whichever comes first based on IMWG criteria for MM participants, based on Lugano criteria for DLBCL participants, and based on IWG response criteria for AML participants.
Expansion Part A: Overall Survival (OS) of GEN3014 | Up to 8 years
  OS is defined as the time from the date of first dose to the date of death due to any cause.
Expansion Part A: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) per CTCAE Version 5.0 | From first dose until the end of the safety follow-up period (30 days after last dose) (Up to 8 years)
Expansion Part A: Number of Participants with Anti-Drug Antibody (ADA) of GEN3014 | From first dose until treatment discontinuation (Up to 8 years)
Expansion Part A: Maximum (peak) Plasma Concentration (Cmax) of GEN3014 | Predose and postdose at multiple timepoints up to Cycle 6 (Cycle length=28 days); Pre-dose and 5 minutes post end of infusion from Cycle 7 and beyond (Up to 8 years)
Expansion Part A: Pre-dose (trough) Concentrations (Ctrough) of GEN3014 | Predose and postdose at multiple timepoints of each Cycle (Cycle length=28 days) (Up to 8 years)
Expansion Part A: Area Under the Concentration Time Curve From Zero to Last Quantifiable Sample (AUC0-last) | Predose and postdose at multiple timepoints up to Cycle 6 (Cycle length=28 days); Pre-dose and 5 minutes post end of infusion from Cycle 7 and beyond (Up to 8 years)
Expansion Part A: Area Under the Concentration Time Curve From Zero to 168 hours (AUC0-168 h) | Predose and postdose at multiple timepoints up to Cycle 6 (Cycle length=28 days); Pre-dose and 5 minutes post end of infusion from Cycle 7 and beyond (Up to 8 years)
Expansion Part B: Ctrough Levels of GEN3014 IV or Daratumumab SC on Cycle 3 Day 1 | Cycle 3 Day 1 (cycle = 28 days)
Expansion Part B: Very Good Partial Response (VGPR), or better of GEN3014 IV vs Daratumumab SC | Up to 8 years
Expansion Part B: Complete Response (CR) or better of GEN3014 IV vs Daratumumab SC | Up to 8 years
Expansion Part B: Duration of Response (DOR) of GEN3014 IV vs Daratumumab SC | Up to 8 years
  DOR is defined as time from first response (PR or better) to time of disease progression or death (due to any cause), whichever comes first based on IMWG criteria for MM participants.
Expansion Part B: Time-to-response (TTR) of GEN3014 IV vs Daratumumab SC | Up to 8 years
  TTR is defined as the time from date of randomization to time of response (PR or better) based on IMWG criteria for MM participants.
Expansion Part B: Progression-free Survival (PFS) of GEN3014 IV vs Daratumumab SC | Up to 8 years
  PFS is defined as the time from date of randomization to the date of progression or death (due to any cause), whichever comes first based on IMWG criteria for MM participants.
Expansion Part B: Overall Survival (OS) of GEN3014 IV vs Daratumumab SC | Up to 8 years
  OS is defined as the time from date of randomization to the date of death due to any cause.
Expansion Part B: Time to Next Therapy (TTNT) | Up to 8 years
  Time to next therapy (TTNT) for participants in the Expansion Part B is defined as the time from date of randomization to the start of subsequent anti-cancer therapy.
Expansion Part B: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) per CTCAE Version 5.0 | From first dose until the end of the safety follow-up period (30 days after last dose) (Up to 8 years)
Expansion Part B: Number of Participants with Anti-Drug Antibody (ADA) of GEN3014 and Anti-daratumumab Antibodies | From first dose until treatment discontinuation (Up to 8 years)

CONTACTS AND LOCATIONS:
Overall Officials: Study Official, Study Director — Genmab
Locations (52):
- United States (3):
  - John Theurer Cancer Center, Hackensack, New Jersey
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Medical college of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Northern Health, Epping
  - The Alfred Hospital, Melbourne
  - Royal Prince Alfred Hospital, Sydney
- Bosnia and Herzegovina (3):
  - University Clinical Center of the Republic of the Srpska, Banja Luka
  - Klinika za hematologiju KCUS, Sarajevo
  - UKC - University Clinical Center Tuzla, Tuzla
- Czechia (5):
  - Fakultni Nemocnice Brno, Brno
  - Vseobecna fakultni nemocnice, New Town
  - Fakultni Nemocnice Hradec Kralove FNHK, Nový Hradec Králové
  - Fakultni Nemocnice Olomouc (FNOL), Olomouc
  - FNO - Fakultni nemocnice Ostrava, Poruba
- Denmark (2):
  - Aalborg Universitet, Aalborg
  - Vejle Hospital, Vejle
- France (2):
  - CHRU de Lille, Lille
  - CHRU de Nantes, Nantes
- ARENSIA Exploratory Medicine LLC, Tbilisi, Georgia
- Greece (4):
  - Alexandra General Hospital, Athens
  - Evangelismos Hospital NKUA, Athens
  - University General Hospital of Patras, Rio
  - Ahepa University General hospital, Thessaloniki
- Szabolcs-Szatmar-Bereg County Hospitals and University Hospital, Josa Andras University Hospital, Nyíregyháza, Hungary
- Malaysia (4):
  - Hospital Ampang, Ampang
  - Hospital Sultanah Aminah, Johor Bahru
  - Hospital Umum Sarawak, Kuching
  - Beacon Hospital, Petaling Jaya
- Institute of Oncology, ARENSIA Exploratory Medicine, Chisinau, Moldova
- Netherlands (3):
  - Maastricht UMC, Maastricht
  - Erasmus MC, Rotterdam
  - UMC Utrecht, Utrecht
- New Zealand (4):
  - Christchurch Hospital, Christchurch
  - Auckland Cancer Trials Centre, Grafton
  - Palmerston North Hospital, Palmerston North
  - North Shore Hospital, Takapuna
- University Clinic of Hematology, Skopje, North Macedonia
- Makati Medical Center, Makati City, Philippines
- Poland (4):
  - University Centrum Kliniczne, Gdansk
  - Pratia Onkologia Katowice, Katowice
  - Pratia MCM, Krakow
  - Wroclaw Medical University, Wroclaw
- South Korea (5):
  - Chonnam National University Hwasun Hospital, Gwangju
  - Pusan National University Hospital PNUH, Pusan
  - Gachon University Gil Medical Center, Seongnam
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
- Spain (2):
  - University of Navarra, Pamplona
  - University Hospital of Salamanca, Salamanca
- Sweden (2):
  - Karolinska Institute, Huddinge
  - Universitetssjukhuset i Lund, Lund
- Arensia Exploratory Medicine, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No